CLINICAL TRIAL: NCT06895369
Title: The Efficacy and Safety of Pucotenlimab Combined With TP Chemotherapy Regimen (Cisplatin and Docetaxel) as Neoadjuvant Therapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: The Efficacy and Safety of Pucotenlimab Combined With TP Chemotherapy as Neoadjuvant Therapy for Locally Advanced HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XiaohuaJiang
Record Dates: First submitted 2025-03-11; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Pucotenlimab; Squamous Cell Carcinoma of Head and Neck; Neoadjuvant Therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Patients will receive 3 cycles of Pucotenlimab combined with TP (cisplatin + docetaxel) as neoadjuvant therapy, followed by standard surgical treatment and postoperative histopathological examination.
  Interventions: Drug: Pucotenlimab

INTERVENTIONS:
Drug: Pucotenlimab — patients will receive 3 cycles of pucotenlimab combined with TP (cisplatin + docetaxel) as neoadjuvant therapy, followed by standard surgical treatment
  Other Names: Cisplatin; Docetaxel

SUMMARY:
Study Objective: To evaluate the efficacy and safety of pucotenlimab combined with TP (cisplatin + docetaxel) as neoadjuvant therapy for locally advanced head and neck squamous cell carcinoma (HNSCC).

Study Design: This is a single-arm interventional study. Intervention: Patients will receive 3 cycles of pucotenlimab combined with TP (cisplatin + docetaxel) as neoadjuvant therapy, followed by standard surgical treatment and postoperative histopathological examination.

Endpoints: Pathological complete response rate (pCR) after surgery, major pathological response rate (MPR) of the treatment regimen, disease-free survival (DFS), and overall survival (OS).

Hypothesis: The combination of pucotenlimab and TP (cisplatin + docetaxel) as neoadjuvant therapy for locally advanced HNSCC is expected to improve pathological response rates and enhance patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 70 years old.
2. Diagnosis: Histopathologically confirmed head and neck squamous cell carcinoma (HNSCC) of the oropharynx, oral cavity, hypopharynx, or larynx, classified as Stage III or IV A according to the AJCC Cancer Staging Manual (8th Edition).
3. Measurable Disease: At least one measurable primary lesion per RECIST 1.1 criteria.
4. Treatment Status: Treatment-naïve patients with no prior therapy for the disease.
5. Performance Status: ECOG performance status of 0-1.
6. Surgical Eligibility: Deemed eligible for elective standard surgery followed by standard adjuvant chemoradiotherapy/radiotherapy, as assessed by the investigator.
7. Autoimmune Disease: No active autoimmune diseases.
8. Concurrent Malignancy: No concurrent malignancies.
9. Life Expectancy: ≥6 months.
10. Biomarker Testing: Available tumor tissue samples for PD-L1 testing via Combined Positive Score (CPS) using 22C3 pharmDx assay (DAKO).
11. Hematologic Parameters:

    * ANC ≥1.5×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥100 g/L, WBC ≥3.5×10⁹/L.
    * No transfusion within 7 days or bleeding tendency.
12. Liver Function: ALT, AST, ALP, and total bilirubin ≤1.5× upper limit of normal (ULN).
13. Renal Function: Serum creatinine ≤1.5× ULN or creatinine clearance >60 mL/min.
14. HPV Status: HPV status confirmed via p16 immunohistochemistry (IHC) and/or in situ hybridization (ISH).
15. Informed Consent: Voluntarily participates and signs informed consent. For participants unable to consent due to incapacity, consent must be provided by a legally authorized representative. For illiterate participants, an impartial witness must attest to the informed consent process.

Exclusion Criteria:

1. Cachexia or multiple organ failure.
2. Active autoimmune disease(s) requiring systemic treatment (excluding vitiligo, resolved childhood asthma/atopy, or controlled hypothyroidism on hormone replacement).
3. Concurrent second primary malignancy (e.g., esophageal cancer).
4. Severe active infection requiring systemic therapy.
5. Uncontrolled comorbid medical conditions that may compromise protocol compliance, per investigator judgment, including:

   * Severe cardiovascular/cerebrovascular diseases,
   * Uncontrolled diabetes/hypertension,
   * Active peptic ulcer,
   * Uncontrolled infections.
6. Dementia, altered mental status, or cognitive impairment affecting informed consent or questionnaire completion.
7. Grade ≥2 peripheral neuropathy (per CTCAE v5.0).
8. Grade ≥2 hearing impairment (per CTCAE v5.0).
9. History of malignancy within the past 5 years (excluding cured non-melanoma skin cancer or carcinoma in situ).
10. Known HIV-positive status or AIDS.
11. Nasopharyngeal carcinoma or squamous cell carcinoma originating outside oral cavity, oropharynx, hypopharynx, or larynx (e.g., sinonasal tract, paranasal sinuses, or unknown primary).
12. Participation in another interventional clinical trial or use of investigational drugs within 30 days prior to screening.
13. Systemic glucocorticoids (>10 mg/day prednisone equivalent) or immunosuppressive agents within 14 days prior to randomization.

    • Exceptions: Inhaled/topical steroids or physiologic replacement doses for adrenal insufficiency.
14. Pregnancy, breastfeeding, or refusal of contraception by subjects of childbearing potential.
15. Active infection requiring treatment or systemic antimicrobial use within 1 week prior to first dose.
16. Live vaccines administered within 30 days before first dose or during the study.
17. Vulnerable populations (e.g., severe psychiatric disorders, cognitive impairment, critically ill patients, prisoners, pregnant individuals).
18. Other conditions deemed by the investigator to preclude safe study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | The anticipated completion date is within 3.5 months after the enrollment of the last patient, with the overall study expected to conclude within 2 years following the enrollment of the first patient.
  Pathological complete response rate (pCR) after surgery

SECONDARY OUTCOMES:
Major pathological response rate | The anticipated completion date is within 3.5 months after the enrollment of the last patient, with the overall study expected to conclude within 2 years following the enrollment of the first patient.
  major pathological response rate (MPR) of the treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Jiang, Master, Study Chair — Sir Run Run Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We have no IPD sharing plan.